CLINICAL TRIAL: NCT03690986
Title: Integrated Pilot Biomarker Trial of VX15/2503 in Combination With Ipilimumab or Nivolumab in Patients With Head and Neck Cancer
Brief Title: VX15/2503 in Combination With Ipilimumab or Nivolumab in Patients With Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Vaccinex Inc. (Industry)
Responsible Party: Principal Investigator, Conor Steuer, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00103534; NCI-2018-01263 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4402-18 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pepinemab; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group A (VX15/2503) (Experimental): Patients receive VX15/2503 IV over 60 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.
  Interventions: Biological: VX15/2503
- Group B (VX15/2503, ipilimumab) (Experimental): Patients receive VX15/2503 IV over 60 minutes and ipilimumab IV over 90 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.
  Interventions: Biological: VX15/2503; Biological: Ipilimumab
- Group C (VX15/2503, nivolumab) (Experimental): Patients receive VX15/2503 IV over 60 minutes and nivolumab IV over 60 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.
  Interventions: Biological: VX15/2503; Biological: Nivolumab
- Group D (nivolumab) (Experimental): Patients receive nivolumab IV over 60 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.
  Interventions: Biological: Nivolumab
- Group E (ipilimumab) (Experimental): Patients receive ipilimumab IV over 90 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.
  Interventions: Biological: Ipilimumab
- Group F (no treatment) (No Intervention): Patients undergo standard of care surgery.

INTERVENTIONS:
Biological: VX15/2503 — Given IV
  Other Names: moAb VX15/2503; Anti-SEMA4D Monoclonal Antibody VX15/2503; Pepinemab
  Arms: Group A (VX15/2503); Group B (VX15/2503, ipilimumab); Group C (VX15/2503, nivolumab)
Biological: Ipilimumab — Given IV
  Other Names: BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Group B (VX15/2503, ipilimumab); Group E (ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Group C (VX15/2503, nivolumab); Group D (nivolumab)

SUMMARY:
This phase I trial studies how well anti-semaphorin 4D (SEMA4D) monoclonal antibody VX15/2503 (VX15/2503) with or without ipilimumab and/or nivolumab work in treating patients with stage I-IVA head and neck squamous cell cancer. Monoclonal antibodies, such as VX15/2503, ipilimumab, and nivolumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To evaluate the effect of VX15/2503 alone and VX15/2503 in combination with immune checkpoint inhibitors, ipilimumab or nivolumab, on the immune profile in the tumor microenvironment and in peripheral blood.

SECONDARY OBJECTIVE:

To extend the previously reported safety profile of single agent VX15/2503 to the combination of VX15/2503 and immune checkpoint inhibitors, ipilimumab or nivolumab, in patients with head and neck squamous cell carcinoma.

OUTLINE: Patients are randomized to 1 of 6 groups.

GROUP A: Patients receive VX15/2503 intravenously (IV) over 60 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.

GROUP B: Patients receive VX15/2503 IV over 60 minutes and ipilimumab IV over 90 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.

GROUP C: Patients receive VX15/2503 IV over 60 minutes and nivolumab IV over 60 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.

GROUP D: Patients receive nivolumab IV over 60 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.

GROUP E: Patients receive ipilimumab IV over 90 minutes on day 1. Beginning days 17-36, patients undergo standard of care surgery.

GROUP F: Patients undergo standard of care surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-IVA cytologically or histologically-proven head and neck squamous cell carcinoma (HNSCC), p16 positive and negative allowed
* Oropharyngeal tumors must have p16 testing done
* Cancer confirmed to be surgically resectable, with surgery evaluation with planned resection
* Archival tissue prior to treatment available from at most 6 months prior to study enrollment. Otherwise new pre-treatment biopsy mandatory
* No prior treatment for HNSCC
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count ≥ 1,500 cells/µL
* Platelets ≥ 100,000/µL
* Hemoglobin ≥ 9.0g/dL (may receive packed red blood cell [prbc] transfusion)
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Albumin ≥ 3.0 g/dL
* Serum creatinine ≤ 1.5 x ULN
* Calculated creatinine clearance of ≤ 50 mL/min
* International normalized ratio (INR) ≤ 1.5. Anticoagulation is allowed only with low molecular weight heparin (LMWH). Patient receiving LMW heparin on stable therapeutic dose for more than 2 weeks or with factor Xa level < 1.1 units/mL (U/mL) are allowed on the trial
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Ability to understand and willingness to sign a written informed consent document
* Female subjects of childbearing potential must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) for the duration of study treatment and 3 months after completion
* Male subjects must agree to use adequate contraception (e.g., condoms; abstinence) for the duration of study treatment and 3 months after completion
* Female subjects of childbearing age must have a negative serum pregnancy test at study entry

Exclusion Criteria:

* Poor venous access for study drug administration
* Nasopharynx cancer, cancer of unknown primary, sinonasal cancer
* Determined not to be a surgical candidate due to medical co-morbidities
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation)
* Prior organ allograft or allogeneic bone marrow transplantation
* Subjects with any active autoimmune disease or history of known or suspected autoimmune disease except for subjects with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Women who are pregnant or lactating
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* Clinical evidence of bleeding diathesis or coagulopathy
* Prior invasive malignancy (except non-melanomatous skin cancer, low or intermediate risk prostate cancer, or in situ carcinoma fully resected) unless disease free for a minimum of one year
* Patients that have had prior treatment for HNSCC are not eligible
* Active bacterial or fungal infections requiring systemic treatment within 7 days of treatment
* Use of other investigational drugs (drugs not marked for any indication) within 28 days or at least 5 half-lives (whichever is longer) before study drug administration
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Non-oncology vaccines within 28 days prior to or after any dose of ipilimumab
* No archival tissue available pre-study treatment, and repeat biopsy not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in immune profile in the tumor microenvironment | Baseline up to 4-8 weeks after surgery
  Specimens from surgical resection will be collected under the guidance of the collaborating pathologist and tissue procurement staff at the time of surgery to capture tissue in excess of that needed for clinical staging and diagnostic purposes. Tumor specimens will be fixed in 10% formalin, embedded in paraffin and biomarkers related to activated HNSCC stroma will be assessed via immunohistochemical analysis.
Change in circulating percentage of immune suppressor subsets in peripheral blood | Baseline up to 4-8 weeks after surgery
  Blood samples will be collected and peripheral blood mononuclear cells will be isolated from these samples and stored in -80°C freezers until analysis. Multi-parameter flow cytometry will be utilized to phenotype immune effector cells. The impact of treatment on the circulating percentage of immune suppressor subsets that may serve as predictors of response to immune checkpoint inhibition. All data will be expressed as the percentage of total circulating peripheral blood cells with each respective phenotype.
Phenotypic shifts in T lymphocyte subsets in peripheral blood | Baseline up to 4-8 weeks after surgery
  Blood samples will be collected and peripheral blood mononuclear cells will be isolated from these samples and stored in -80°C freezers until analysis. Blood will be analyzed by multi-parameter flow cytometry to identify systemic phenotypic shifts mediated by VX15/2503 in combination with immune checkpoint inhibition.

SECONDARY OUTCOMES:
Incidence of adverse events assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 4-8 weeks after surgery
  Adverse events will be classified using MedDRA System Organ Classes and Preferred Terms. Furthermore, serious adverse events, adverse events (AEs) with a severity grade of 3 or above using NCI CTCAE version 4.0, AEs deemed related to study drug, AEs leading to discontinuation of study drug, and AEs leading to death will also be summarized in preferred term by system organ class and listed on an individual subject basis.

CONTACTS AND LOCATIONS:
Overall Officials: Conor Steuer, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States